CLINICAL TRIAL: NCT01370720
Title: Effect of the Oral Administration in IBS Patients of the Association of 200 mg Micronised Palmitoylethanolamide (PEA) and 20 mg Polydatin, on Parameters of Intestinal Inflammation and Visceral Hyperalgesia.
Brief Title: Safety and Efficacy Study of PEA and Polydatin on Intestinal Inflammation and Visceral Hyperalgesia in IBS Patients
Acronym: CMD-IBS09(2)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MARIA CRISTINA COMELLI (Industry)
Responsible Party: Sponsor-Investigator, MARIA CRISTINA COMELLI, Head,R&D, CM&D Pharma Limited
Organization: CM&D Pharma Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CM&D Pharma Limited
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; mast cell activation; low grade inflammation; visceral hyperalgesia
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recoclix (CM&D Pharma Limited) (Active Comparator): Recoclix: two tablets per day for 12 weeks
  Interventions: Dietary Supplement: Recoclix
- Placebo (Placebo Comparator): IBS patients
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Recoclix — tablets; 200 mg PEA+20 mg polydatin; 2 tablets/day; 12 weeks
  Arms: Recoclix (CM&D Pharma Limited)
Other: Placebo — tablets, 2tablets/day, 12 weeks
  Arms: Placebo

SUMMARY:
Despite the pathophysiology of IBS remains largely unsettled, several mechanisms have been proposed to explain symptom generation. These include psychosocial factors, altered gastrointestinal motor function and altered perception of visceral stimuli because of chronic low-grade inflammation and increased nociceptive mediator release by inflammatory cells, particularly mast cells.

The aim of this pilot study is to provide evidence of:

1. intestinal mast cell (MC) infiltration and activation in IBS patients;
2. down-modulation of MC activation by the oral administration of the association of palmitoylethanolamide (PEA) and polydatin in IBS patients.

DETAILED DESCRIPTION:
The number of inflammatory cells in the gut wall of IBS patients is increased in comparison to asymptomatic controls. A significant increase in the number of both mast cells and T-lymphocytes in the mucosa of IBS patients have been reported. Electron microscopic studies demonstrated that mast cells were more frequently degranulated in IBS, suggesting their increased state of activation. Accordingly, an increased mucosal release of preformed mediators, such as histamine and tryptase, as well as de novo synthesis and secretion of arachidonic acid end products (e.g. prostaglandin E2) have been demonstrated. These mediators are known to target sensory nerve pathways, including those innervating the gastrointestinal tract, leading to visceral hyperalgesia.

Electron microscopic studies showed that the mean distance between inflammatory cells and enteric nerves is significantly reduced in IBS patients, thus providing a conceptual basis for a putative pathogenetic role of low-grade inflammation on sensory-motor dysfunction in IBS. Activated mast cells in close proximity to mucosal colonic innervation correlated with the frequency and severity of abdominal pain. Evidence that mast cell mediators of IBS patients, but not controls, evoked activation of nociceptive sensory afferent neurons are available, thus providing a possible mechanism through which mast cells can evoke pain in IBS patients. Similar results has been recently reported following the administration into the rat colon of supernatants collected from human IBS colonic biopsy samples in culture. This nociceptive effect on murine sensory neurons was inhibited by serine protease inhibitors and a Protease Activating Receptor-2 antagonist.

ELIGIBILITY:
Inclusion Criteria:

* IBS patients (both males and females) with positive diagnosis based on Rome III criteria (all IBS subtypes will be included)
* Age in the range 18-70 years
* Subjects capable of conforming to the study protocol
* Subjects who have given their free and informed consent

Exclusion Criteria:

* Any relevant organic, systemic or metabolic disease, such as celiac disease, IDDM (Insulin-Dependant Diabetes Mellitus), Insulin-Independent Diabetes Mellitus, metabolic syndrome, pelvic organ prolapse, and urinary incontinence.
* Subjects with ascertained intestinal organic diseases (ulcerative colitis, Crohn's disease, microscopic colitis, infectious colitis, ischemic colitis, complicated diverticular disease).
* Subjects with untreated food intolerance, i.e. remaining symptomatic despite the withdrawal of the suspected food
* Previous major abdominal surgeries
* Females of childbearing potential, in the absence of effective contraceptive methods
* Subjects who become unable to conform to protocol
* Subjects who are continuously taking contact laxatives
* Subjects who have been continuously administered glucocorticoids, anti-histaminergic and mast cell stabilizer drugs within the previous 30 days
* Subjects who have been continuously administered trimebutine within the previous 30 days
* Treatment with any investigational drug within the previous 30 days
* Recent history or suspicion of alcohol abuse or drug addiction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Changes from screening visit of mast cell infiltration and activation in biopsy samples of colon mucosa from IBS patients, following 12 weeks of dietary supplementation with palmitoylethanolamide (PEA) and polydatin | screening visit and after 12 weeks
  Comparison between healthy volunteers and IBS patients (screening visit) on the following parameters:
  * number of infiltrating mast cells (ICH)
  * mast cell activation, as per histamine and tryptase release in the surnatant of cultured colon biopsy samples
  Comparison between active and placebo supplemented IBS patients (after 12 weeks from randomization) on the following parameters:
  * number of infiltrating mast cells (ICH)
  * mast cell activation, as per histamine and tryptase release in the surnatant of cultured colon biopsy samples

SECONDARY OUTCOMES:
Changes in biomarkers related to the endocannabinoid system | 12 weeks after randomization
  Comparison between active and placebo supplemented IBS patients (after 12 weeks from randomization) on the level of anandamide, 2-AG, PEA, CB1, CB2, FAAH (LC-APCI-MS; immunoblotting)
Changes from screening visit of other inflammatory cell subsets in biopsy samples of colon mucosa from IBS patients, following 12 weeks of dietary supplementation with palmitoylethanolamide (PEA) and polydatin | screening visit and after 12 weeks
  Comparison between active and placebo supplemented IBS patients (after 12 weeks from randomization) of the number of other inflammatory cell subsets (ICH)
Safety assessment by no changes in laboratory parameters and vital signs | 4, 8, 12 weeks after randomization
  * Laboratory test (blood cell count, AST, ALT, creatinine, gamma-GT, alkaline phosphatase, total bilirubin, glucose, N, Na, K, Ca)
  * Physical examination and vital signs (systolyc and diastolic blood pressure, heart rate, respiratory rate)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept Internal Medicine and Gastroenterology, Policlinico Sant'Orsola-Malpighi, Bologna, Italy

REFERENCES:
- [Derived] Cremon C, Stanghellini V, Barbaro MR, Cogliandro RF, Bellacosa L, Santos J, Vicario M, Pigrau M, Alonso Cotoner C, Lobo B, Azpiroz F, Bruley des Varannes S, Neunlist M, DeFilippis D, Iuvone T, Petrosino S, Di Marzo V, Barbara G. Randomised clinical trial: the analgesic properties of dietary supplementation with palmitoylethanolamide and polydatin in irritable bowel syndrome. Aliment Pharmacol Ther. 2017 Apr;45(7):909-922. doi: 10.1111/apt.13958. Epub 2017 Feb 6. PMID 28164346